CLINICAL TRIAL: NCT00714038
Title: CARE - Quality Development in Asthma in General Practice
Brief Title: CARE - Quality Improvement in Asthma Secondary Prevention in Primary Care, Through Delegation of Consultations to the Nurse.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-RDK-DUM-2008/1
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Asthma
Keywords: Quality development project; primary care nurses; asthma; patient compliance; follow-up
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with asthma in primary care

SUMMARY:
Quality Improvement in Primary Care: delegation of check-ups to nurses in general practice

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with asthma

Exclusion Criteria:

* patients with copd

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2122 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Lung function, improvements in lung function over time, patient compliance with treatment | baseline, when necessary and at 1 year control

SECONDARY OUTCOMES:
Number of visits per patient, drop-out rate | annually

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Ommen, MD, Study Chair — Lægerne i Løgumkloster I/S, Denmark; Dorte Knudsen, Study Chair — Lægerne Sønderåparken, Denmark
Locations (93):
- Denmark (93):
  - Research Site, Aabenraa
  - Research Site, Aabybro
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Albertslund
  - Research Site, Arhus C
  - Research Site, Arhus N
  - Research Site, Ballerup Municipality
  - Research Site, Birkerød
  - Research Site, Brabrand
  - Research Site, Bryrup
  - Research Site, Brønshøj
  - Research Site, Christiansfeld
  - Research Site, Dybvad
  - Research Site, Elsinore
  - Research Site, Erslev
  - Research Site, Espergorde
  - Research Site, Fakse
  - Research Site, Fredericia
  - Research Site, Frederikshavn
  - Research Site, Frostruo
  - Research Site, Gedsted
  - Research Site, Gram
  - Research Site, Haderslev
  - Research Site, Hadsund
  - Research Site, Hasselager
  - Research Site, Hedehusene
  - Research Site, Herfølge
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Hinnerup
  - Research Site, Hjørring
  - Research Site, Hobro
  - Research Site, Holbæk
  - Research Site, Holstebro
  - Research Site, Holte
  - Research Site, Horsens
  - Research Site, Humlaek
  - Research Site, Hurup Thy
  - Research Site, Højer
  - Research Site, Hørning
  - Research Site, Hørsholm
  - Research Site, Ikast
  - Research Site, Jægerspris
  - Research Site, Karlslunde
  - Research Site, Karup
  - Research Site, Kåstrup
  - Research Site, Kbh. NV
  - Research Site, Kerteminde
  - Research Site, Kjellerup
  - Research Site, Kolding
  - Research Site, Kongens Lyngby
  - Research Site, København S
  - Research Site, Køge
  - Research Site, Låsby
  - Research Site, Lemvig
  - Research Site, Middelfart
  - Research Site, Møldrup
  - Research Site, Nordborg
  - Research Site, Nyborg
  - Research Site, Nykobing Sj�lland
  - Research Site, Nykøbing Falster
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Randers
  - Research Site, Ribe
  - Research Site, Roskilde
  - Research Site, Rødovre Municipality
  - Research Site, Sakskøbing
  - Research Site, Silkeborg
  - Research Site, Skive
  - Research Site, Skovlunde
  - Research Site, Skørping
  - Research Site, Slagelse
  - Research Site, Slangerup
  - Research Site, Snekkersten
  - Research Site, Solbjerg
  - Research Site, Solrod Srand
  - Research Site, Storvorde
  - Research Site, Støvring
  - Research Site, Svendborg
  - Research Site, Sønderborg
  - Research Site, Tarm
  - Research Site, Terndrup
  - Research Site, Thisted
  - Research Site, Uldum
  - Research Site, Vallensaek Strand
  - Research Site, Vanløse
  - Research Site, Varde
  - Research Site, Vejle
  - Research Site, Viborg
  - Research Site, Virum
  - Research Site, Vojens